CLINICAL TRIAL: NCT03208673
Title: Optive Brand For Day And Night Dry Eye Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMO-EAME-EYE-0485
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Optive® Fusion + Optive® Gel Drop (Experimental): Optive® Fusion eyedrop will be used as needed up to four times a day but at least twice a day. The eyedrop will be used once in the evening; the gel drop being instilled any time during the last hour prior to sleep. The treatment regimen will be used for one month.
  Interventions: Device: Optive® Fusion + Optive® Gel Drop

INTERVENTIONS:
Device: Optive® Fusion + Optive® Gel Drop — Optive® Fusion eyedrop will be used as needed up to four times a day but at least twice a day. The eyedrop will be used once in the evening; the gel drop being instilled any time during the last hour prior to sleep.

SUMMARY:
This is an open label study of Optive eyedrops and gel combination for day and night dry eye management

ELIGIBILITY:
Inclusion Criteria:

* OSDI score of ≥ 23
* Ocular comfort at waking <65 on 100-point scale
* Conjunctival staining Grade ≥ 2 (scale 0 to 4) in at least one eye
* Use of eyedrops for the relief of dry eye symptoms for at least one month
* Best corrected visual acuity in each eye of at least 20/25
* Have normal eyes with the exception of the need for visual correction; subjects must be willing to cease contact lens wear for the duration of the study
* Be willing and able to adhere to the instructions set in the clinical protocol and maintain the appointment schedule

Exclusion Criteria:

* Use of Benzalkonium Chloride (BAK) preserved eyedrops in the last month
* Use of Optive brand eyedrops in the last month
* Monocular participants (only one eye with functional vision).
* Contact lens wear during the study
* History of herpetic keratitis, ocular surgery or irregular cornea;
* Known pregnancy or lactation during the study period
* Participation in any clinical trial within 30 days of the enrollment visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameena Haque, Study Director — Allergan
Locations (1):
- Ocular Technology Group - international, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Optive® Fusion™ and Optive® Gel Drop: A CE marked eyedrop, containing 0.1% sodium hyaluronate, 0.5% carmellose sodium and 0.9% glycerol for daytime use. The eyedrop will be used as needed up to four times a day but at least twice a day and A CE marked gel, containing 0.5% carboxymethylcellulose sodium and 0.9% glycerol for night time use. The eyedrop will be used once in the evening; the gel drop being instilled any time during the last hour prior to sleep.
Period: Overall Study
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
Number analyzed (Participants) | 32
Age, Continuous [Mean (Full Range); unit: Years] | 52.13 [33 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data not collected for these data points.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Disease Index (OSDI) Total Score
Description: A 12-question survey used to measure the symptoms of dry eye disease. Each of the 12 individual questions rate one symptom on a 0-4 scale, with 4 meaning that the symptom is present all of the time and 0 meaning the symptom is present none of the time. The overall ODSI score is calculated by adding all of the values from the 12 questions, multiplying that value by 25, and dividing the resulting value by the number of questions answered. This results in an overall scale that ranges from 0-100, with 100 being severe dry eye symptoms and 0 being no dry eye symptoms.
Time Frame: Change from baseline to (day 30 +/- 3 days)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
Number analyzed (Participants) | 32
Scores on a scale | -12.85 (14.80)
Statistical Analysis 1: Comparison: Optive® Fusion™ and Optive® Gel Drop; Test type: Superiority; p = .001, t-test, 2 sided; Ratio of Geometric mean = 0.5628, 95% CI 2-sided [0.4395 to 0.7204]

2. Primary Outcome: Measured Lissamine Green Bulbar Conjunctival Staining (mm2)
Description: The Lissamine Green (LG) bulbar conjunctival staining was analysed post-hoc for both eyes. The photos were masked and for each image the Staining Area was measured (mm2).
Time Frame: Change from baseline to (day 30 +/- 3 days)
Measure: Mean (Standard Deviation); unit: mm2
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
Number analyzed (Participants) | 32
mm2
  Nasal | 0.03 (0.04)
  Temporal | 0.03 (0.08)
Statistical Analysis 1: Comparison: Optive® Fusion™ and Optive® Gel Drop; Nasal; Test type: Superiority; p = 0.025, t-test, 1 sided
Statistical Analysis 2: Comparison: Optive® Fusion™ and Optive® Gel Drop; Temporal; Test type: Superiority; p = 0.312, t-test, 1 sided

3. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS): Symptomatology Upon Waking
Description: The participant rated the severity of their symptomatology upon waking using a VAS scale. Participants put a mark on a 100 millimeter line where 0 (far left on the line) = no symptoms to 100 (far right on the line) = most severe symptoms.
Time Frame: Baseline (day 0) to (day 30 +/- 3 days)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
Number analyzed (Participants) | 32
scores on a scale
  Comfort at Baseline | 30.22 (17.96)
  Comfort at Day 30 | 58.02 (29.56)
  Dry at Baseline | 59.08 (27.34)
  Dry at Day 30 | 42.28 (32.74)
  Gritty at Baseline | 52.95 (27.43)
  Gritty at Day 30 | 31.09 (31.81)
  Vision at Baseline | 49.00 (30.91)
  Vision at Day 30 | 64.84 (29.98)
Statistical Analysis 1: Comparison: Optive® Fusion™ and Optive® Gel Drop; Comfort; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 2: Comparison: Optive® Fusion™ and Optive® Gel Drop; Dry; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 3: Comparison: Optive® Fusion™ and Optive® Gel Drop; Gritty; Test type: Superiority; p < 0.001, t-test, 1 sided
Statistical Analysis 4: Comparison: Optive® Fusion™ and Optive® Gel Drop; Vision; Test type: Superiority; p < 0.001, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Baseline (day 0) to (day 30 +/- 3 days)
Description: Did not meet 5% threshold
Arm/Group | Optive® Fusion™ and Optive® Gel Drop
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

(Note that this agreement language may appear in the study protocol)

DOCUMENTS (2):
  • Study Protocol (2017-05-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT03208673/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT03208673/SAP_001.pdf